CLINICAL TRIAL: NCT06690528
Title: Conversion Surgery Vs. Palliative Care in Pancreatic Cancer Oligometastatic to the Liver (SONAR: Surgery in Oligometastatic PaNcreatic CAnceR) a Randomized Controlled Trial
Brief Title: Conversion Surgery Vs. Palliative Care in Pancreatic Cancer Oligometastatic to the Liver
Acronym: SONAR
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Azienda Ospedaliera di Padova (Other)
Collaborators: University of Padova (Other)
Responsible Party: Principal Investigator, Prof. Umberto Cillo, Chief of General Surgery 2 Department - HBP and liver transplantion unit, Azienda Ospedaliera di Padova
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: University of Padova, Italy; 23170 (Other: CET area centro-est Veneto)
Record Dates: First submitted 2024-11-06; First posted 2024-11-15 (Actual); Last update posted 2024-11-15 (Actual); Status verified 2024-11

CONDITIONS: Pancreatic Cancer Metastatic
Keywords: Pancreatic Cancer Metastatic to Liver; Pancreatic Cancer Oligometastatic to Liver; Coversion Surgery Pancreatic Cancer; NEoadiuvant Therapy for Oligometastatic Pancreatic Cancer; Resectable Pancreatic Cancer; Resectable Liver Metastasis in Pancreatic Cancer; Combined Surgery for Metastatic Pancreatic Cancer

STUDY DESIGN:
Intervention Model Description: This is a phase-2 multicenter randomized controlled trial with a 1:1 allocation ratio. Eligible patients with pancreatic cancer oligometastatic to the liver with response/stability after first-line chemotherapy will receive surgical resection or observation/continued chemotherapy. The study will be conducted at different international referral centers with high expertise in pancreatic cancer treatment to ensure the highest standards of quality and an adequate sample size. After the enrollment of the first 20 cases, an independent data monitoring committee (IDMC) will review safety and futility (using 90 days major morbidity + mortality as the endpoint), to allow for early study termination or modification if necessary.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Surgical Resection Arm (Experimental): Patients in this arm will undergo surgical resection of both the primary tumor and liver metastases. The surgical approach, extent of resection, and perioperative management will follow the standard protocols at each participating center. Venous vascular resections might be performed to reach radicality. Either standard or parenchyma sparing liver resections might be performed for resection of the liver metastases. Alternatively, needle ablation/microwave on the liver lesions is possible for lesions <20 mm if technically feasible. Post-operative chemotherapy and/or radiotherapy could be administered as per multi-disciplinary decision based on case-by-case evaluation.
  Interventions: Procedure: Surgical resection of both the primary tumor and liver metastases
- Palliative care arm (No Intervention): Patients in this arm will continue to be treated following palliative care, consisting in observation or continuation of chemotherapy according to investigator's choice and duration of first-line chemotherapy. If required, they will continue with systemic chemotherapy, as received during the initial treatment phase, with a chemotherapy protocol based on the Institution's approved guidelines and adjusted as for clinician's choice.

INTERVENTIONS:
Procedure: Surgical resection of both the primary tumor and liver metastases — Surgical resection of both the primary tumor and liver metastases. The surgical approach, extent of resection, and perioperative management will follow the standard protocols at each participating center. Venous vascular resections might be performed to reach radicality. Either standard or parenchyma sparing liver resections might be performed for resection of the liver metastases. Alternatively, needle ablation/microwave on the liver lesions is possible for lesions <20 mm if technically feasible. Post-operative chemotherapy and/or radiotherapy could be administered as per multi-disciplinary decision based on case-by-case evaluation.
  Arms: Surgical Resection Arm

SUMMARY:
This study investigates the impact of surgical resection compared to palliative care in patients with oligometastatic pancreatic cancer limited to the liver. Specifically, it examines whether surgery after stable disease or response to chemotherapy can improve survival and quality of life. The international, multicenter randomized trial will recruit 56 patients, assigning them to either surgical resection (including tumor and liver metastases) or ongoing palliative care with chemotherapy. Stratification by performance status, tumor markers, and tumor location will ensure balanced study groups. Outcome assessments, conducted over a minimum two-year follow-up, include clinical evaluations, imaging, and quality-of-life metric

DETAILED DESCRIPTION:
Pancreatic cancer is a highly aggressive disease, with advanced-stage diagnosis being the most common presentation, where surgery is usually contraindicated regardless of the number and location of metastases. Among the various metastatic sites, liver involvement is particularly common. The conventional approach for metastatic disease is systemic chemotherapy, aimed at controlling tumor growth, reducing symptoms, and improving quality of life. However, the role of aggressive local therapies, such as surgical removal of the primary tumor and liver metastases, is under active investigation and clinical debate for patients who show response or disease stability following chemotherapy treatment in the context of oligometastatic disease. The oligometastatic stage, defined as the presence of a limited number of metastatic lesions in specific organs, offers a potential opportunity for locoregional interventions. Proponents of surgical intervention argue that complete removal of the tumor following optimal first-line systemic therapy may eradicate the primary cancer source and eliminate or control metastatic sites. This approach could potentially improve disease control, survival, and quality of life for selected patients. This prospective study thus aims to compare the efficacy and safety of a surgical approach versus palliative treatment alone in patients with resectable oligometastatic pancreatic cancer to the liver, with stable disease or therapeutic response following first-line chemotherapy.

This is an international multicenter randomized controlled trial promoted by the University of Padua. The study aims to enroll 28 patients per arm, for a total of 56. The study will include adult patients aged 18 years or older with cytologically or histologically confirmed pancreatic adenocarcinoma and radiologically documented liver metastases. Eligible patients must present with synchronous oligometastatic disease, defined as a limited number of liver metastases (up to 3 lesions) without evidence of extrahepatic metastases, based on a multidisciplinary discussion. The primary pancreatic tumor must still be present at the time of enrollment. Enrolled patients must have received at least 6 months of systemic chemotherapy. Eligible patients with response/stability after first-line chemotherapy will undergo either surgical resection or continuous chemotherapy, depending on the arm to which they are randomized. Patients will be assigned in a 1:1 ratio to either the surgical resection arm (n=28) or the palliative care arm (n=28). Randomization will be performed centrally using a computer-generated randomization sequence. Stratification factors, such as ECOG Performance Status, serum Ca 19-9 level at enrollment, primary pancreatic tumor location, and participating center, will be used to ensure balance between the two study arms. Due to the nature of the interventions, it is not feasible to blind patients and treating physicians to treatment allocation. Upon enrollment, the patient must consent to participate in the above-described randomized study. The two randomization arms are as follows:

A) Surgical Resection Arm: Patients in this arm will undergo surgical resection of both the primary tumor and liver metastases. The surgical approach, extent of resection, and perioperative management will follow the standard protocols of each participating center. Venous vascular resections may be performed to achieve oncologic radicality. Standard or parenchyma-sparing liver resections may be conducted for the resection of liver metastases. Alternatively, percutaneous or microwave ablation of liver lesions <20 mm is possible if technically feasible. Postoperative chemotherapy and/or radiotherapy may be administered based on multidisciplinary decisions and individual case evaluations.

B) Palliative Care Arm: Patients in this arm will continue to receive palliative care, consisting of observation or continuation of chemotherapy based on the investigator's choice and the duration of first-line chemotherapy. If necessary, they will continue with systemic chemotherapy, as received during the initial treatment phase, following an institution-approved chemotherapy protocol adapted to the attending physician's preference. Patients will undergo regular evaluations at predefined intervals throughout the study period. These evaluations will include clinical assessments, laboratory tests, radiologic imaging (such as abdominal and chest CT scans with contrast), quality-of-life assessments, and nutritional evaluations. The frequency of evaluations may vary depending on the study phase but will generally occur every 8-12 weeks according to clinical practice. These assessments will provide data on primary and secondary endpoints. The minimum follow-up specified by the study protocol is 2 years from randomization.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients aged ≥18 years and ≤75 years (at diagnosis).
* Cytologically or histologically confirmed pancreatic adenocarcinoma either resectable or borderline resectable (at diagnosis) according to National Comprehensive Cancer Network (NCCN)4 (see section 5).
* Synchronous oligometastatic disease (at diagnosis), defined as a limited number of radiologically documented liver metastases (up to 3 lesions).
* No evidence of extrahepatic metastases (at diagnosis.)
* Eastern Cooperative Oncology Group (ECOG) performance status (PS) 0-1 (at enrollment)
* Partial response or stable disease after completion of first-line chemotherapy, as determined by RECIST 1.1 criteria21 (modified to exclude any % of increase in the sum of diameters of target lesions) (at enrollment).
* Decreasing or stable (defined as ≤20% increase) serum CA19-9 level after chemotherapy (at enrollment).
* Liver metastases considered resectable (see section 5) or alternatively treatable by needle ablation/microwave once no larger than 20 mm (at enrollment).

Exclusion Criteria:

* Locally advanced pancreatic cancer according to NCCN4.
* Unresectable liver disease (according to multidisciplinary discussion).
* Involvement of other organs.
* Presence of significant comorbidities precluding surgery.
* Pregnancy.
* Contraindications to surgical resection.
* Prior surgical resection of the primary tumor or liver metastases.
* Evidence of extrahepatic metastases.
* Inability to provide informed consent or participate in follow-up assessments.
* Disease progression as determined by RECIST 1.1 criteria21 (modified to include any % of increase in the sum of diameters of target lesions) after chemotherapy.
* Serum CA19-9 level increase >20% after chemotherapy.

Note: Additional specific exclusion criteria may be defined at each participating center based on their institutional guidelines and patient population.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 56 (Estimated)
Dates: Start 2024-11-06 (Actual); Primary Completion 2028-11 (Estimated); Study Completion 2028-11 (Estimated)

PRIMARY OUTCOMES:
Two-year OS (2y-OS) rate | 2 years from randomization.
  The percentage of patients alive after 2 years from randomization.

SECONDARY OUTCOMES:
Progression Free Survival (PFS) | From date of randomization until the date of first documented progression or date of death from any cause, whichever came first, assessed up to 2 years
  The time between randomization and diagnosis of progressive disease.
Surgical mortality and morbidity | 90 days after surgery.
  Surgical mortality and morbidity, graded according to Clavien-Dindo classification, at 90-days after surgery.
Cancer Quality of Life (CQoL) | From date of randomization up to 2 years. The frequency of evaluations may vary depending on the study phase it will generally occur every 8-12 weeks according to clinical practice.
  The EORTC QLQ-C30 is a quality-of-life assessment tool for cancer patients, comprising 30 items that cover physical, emotional, and social aspects of well-being. It includes 15 scales: 5 functional (physical, role, cognitive, emotional, social), 3 symptom (fatigue, nausea/vomiting, pain), 6 single-item symptoms (dyspnea, insomnia, appetite loss, constipation, diarrhea, financial impact), and 1 global health scale. Responses use a scale from 1 to 4, except the global health scale, which ranges from 1 to 7. Scores are transformed to a 0-100 scale; for functional scales, higher scores mean better function, while in symptom scales, higher scores indicate more severe symptoms. This scoring enables monitoring of patient well-being and the impact of treatments.
Pancreatic Cancer Quality of Life (PQoL) | From date of randomization up to 2 years. The frequency of evaluations may vary depending on the study phase it will generally occur every 8-12 weeks according to clinical practice.
  The EORTC QLQ-PAN26 is a quality-of-life assessment tool specifically developed for patients with pancreatic cancer, used alongside the core QLQ-C30 questionnaire. It includes 26 items focused on pancreatic cancer-related symptoms and treatment effects, covering domains such as pain, gastrointestinal symptoms, dietary changes, and emotional issues unique to this patient group. Scales include specific areas like pancreatic pain, digestive issues, altered bowel habits, and jaundice, as well as treatment side effects. Responses follow a 1 to 4 scale, with scores transformed to a 0-100 range; higher scores on symptom scales reflect more severe symptoms, while higher functional scale scores indicate better functioning. This questionnaire allows for targeted monitoring of pancreatic cancer patients' unique challenges and treatment impacts
Treatment-related Adverse Event | From date of randomization up to 2 years.
  Monitoring and documenting adverse events are essential for assessing the safety and tolerability of a treatment, as they help identify and quantify the potential risks associated with the therapy under investigation.

CONTACTS AND LOCATIONS:
Overall Officials: Giovanni Marchegiani, MD, PhD, Professor, Study Chair — University of Padova; Umberto Cillo, Director, MD, Professor, Principal Investigator — University of Padova
Locations (1):
- UOC Chirurgia Generale 2, Azienda Ospedale di Padova, Padua, Italy, Italy

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Guastella R, Perri G, Bassi D, Canitano N, Padoan V, Grandi S, Pellegrini R, Procaccio L, Bergamo F, Lonardi S, Carandina R, Gringeri E, Marchegiani G, Cillo U. Conversion surgery vs. standard of care in pancreaTic cancer oligometastatic to the liver (SONAR: Surgery in Oligometastatic paNcreatic cAnceR) a randomized controlled trial. BMC Cancer. 2026 Jan 12;26(1):44. doi: 10.1186/s12885-025-15183-9. PMID 41526867